Title: Comparison of Etomidate Plus Propofol, Etomidate Alone on Induction of Anesthesia

NCT03820388

Document Date: September 26, 2017

## Statistical Analysis

Sample size calculations were based on our pilot study, and we found MAP to be 80.1 (±10.3) mmHg, 90.3 (±10.4) mmHg, 91.0 (±11.6) mmHg in group P, PE and E at induction. Using PASS 15.0 software, a sample size of 20 patients per group would be needed to detect statistically significant differences with the power of 0.9 and the alpha level of 0.05. Considering a possible 20% dropout rate, 25 patients per group were recruited for the study.

Parametric values were expressed as mean (SD), or percentages of the total number of patients (%). Categorical data were analyzed using  $\chi^2$  or Fisher's exact test as appropriate. The hemodynamic parameters among the three groups were compared using the general linear model (GLM). We also considered time of evaluation as a within-subject factor, and the intervention state as a between-subject factor. The time groups (interaction terms) were considered group differences among the three groups in their responses over time. We used Mauchly's sphericity test for compound symmetry assumption. Differences in hemodynamic variables between the three groups at different time points were compared by post hoc Bonferroni test. P<0.05 was considered statistically significant. All statistical analyses were performed with SPSS 22.0 (SPSS; Chicago, IL, USA).